CLINICAL TRIAL: NCT03115307
Title: A Protocol for a Randomized, Controlled Study to Compare the Use of Gonodotropin-releasing Hormone Agonist Triptoreline (Gonapeptyl®) for Luteal Phase Support Versus Natural Luteal Phase in the Insemination Cycles
Brief Title: Luteal Phase Support in Insemination Cycles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R16171M; 2016-002321-11 (EudraCT Number)
Record Dates: First submitted 2016-11-17; First posted 2017-04-14 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-10

CONDITIONS: Infertility, Female
Keywords: Insemination; Luteal phase support; Gonadotropin-releasing hormone agonist; Triptorelin
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gonapeptyl (Experimental): In the intervention group the patient will get the advice to using triptorelin (Gonapeptyl®) in the eight day after the injection of hCG (Pregnyl®) in the insemination cycle.
  Interventions: Drug: Triptorelin
- Control group (No Intervention): In the control group, there are no luteal phase medications in the insemination cycle.

INTERVENTIONS:
Drug: Triptorelin — Triptorelin 0,1mg/ml subcutaneously once in a luteal phase in insemination cycles.
  Arms: Gonapeptyl

SUMMARY:
This study is a prospective randomized trial with 242 IUI cycles. Patients are randomized in two groups including 121 cycles in each group. A total of 255 cycles in 167 patients are finally recruited. In the first group, the patients will be treated with triptorelin (Gonapeptyl®) in their luteal phase. As for the other group, the patients will undergo the luteal phase without any supportive medication. This study is going to clarify the role of the gonadotropin agonist (triptorelin acetate, Gonapeptyl®) as a luteal phase supporter. The benefit of the treatment is measured by the numbers in the live birth and clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with ovarian stimulation cycles preparing to insemination
* Patients with medical ovarian stimulation protocols including GnRH agonist, aromatase inhibitors and different combinations of GnRH agonists and aromatase inhibitors are included
* Patient's willingness to participate in the study

Exclusion Criteria:

* - Failure in the ovarian stimulation cycle
* Failures in executing the insemination
* Failures in giving the sperm sample
* Major troubles in sperm parameters leading to an inadequate sample to accomplish intrauterine insemination
* Patients with primarily planned progesterone luteal support

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Live birth rate | At possible delivery (about 40 weeks)

SECONDARY OUTCOMES:
Ongoing pregnancy rate | After two weeks
Miscarriage rate | During subsequent about 40 weeks of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Helena Tinkanen, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland